CLINICAL TRIAL: NCT04125225
Title: An Interpretative Phenomenological Analysis of 'Recovery' Following Complete Cytoreductive Surgery.
Brief Title: What Are the Experiences of Patients With Pseudomyxoma Peritonei?
Status: Withdrawn | Type: Observational
Why Stopped: No participants enrolled.
Sponsor: University of Southampton (Other)
Collaborators: Hampshire Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Samuel Downes, Clinical Doctoral Research Fellowship, University of Southampton
Other Study IDs: ERGO ID: 49443; 231042 (Other: IRAS)
Record Dates: First submitted 2019-10-10; First posted 2019-10-14 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Pseudomyxoma Peritonei; Cytoreductive Surgery; Recovery
MeSH Terms: conditions — Pseudomyxoma Peritonei

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Complete cytoreductive surgery (CCRS) is an extensive, and potentially curative, procedure utilised for peritoneal malignancies including Pseudomyxoma peritonei (PMP). This study aims to provide a nuanced understanding of the lived experience of recovery following CCRS over time, with the view to inform future supportive measures for CCRS patients in particular. This study also provides the opportunity to longitudinally examine patient perceptions of 'recovery' in the context of major illness and/or treatment; i.e. what it is to experience recovery, what is important during recovery, perhaps how this changes over time, and what it is to be 'recovered', if this is possible. A greater understanding of the term may have implications in how it is used, or how patients following major illness are approached by healthcare professionals.

Interpretive Phenomenological Analysis (IPA) will be utilised as the guiding methodology in order to answer the study objectives. Potential participants will be approached by the clinical nurse specialist (CNS) involved in the patient's care, and will be offered a 'research study pack', containing a participant information sheet (PIS). A maximum of ten consenting participants will be interviewed on up to six occasions (although only five are planned) across a timeframe of little more than a year, both before and after their surgery. Interviews may take place face-to-face, or via telephone. Data analysis will involve a cyclical process of identifying patterns within the interview transcripts of each participant at each time point, across time points, and between participants. This design will provide an effective means of gathering and analysing rich data from each participant, thus affording a comprehensive insight into the meanings that participants attribute over time to their recovery following CCRS.

This study has been devised in partial fulfilment of a doctorate degree at the University of Southampton.

DETAILED DESCRIPTION:
Complete cytoreductive surgery (CCRS), an extensive procedure increasingly used to treat, and potentially cure, advanced cancers of the peritoneal cavity, including Pseudomyxoma Peritonei (PMP). In a process that can last fourteen hours a typically sizeable number of peritoneal organs or tissues (upon which cancerous cells present) are targeted for tumour nodule removal, or are resected or excised. CCRS is concluded by the administration of hyperthermic intraperitoneal chemotherapy (HIPEC), a warm chemotherapy solution which is gyrated across the peritoneal cavity for one to two hours.

Despite the magnitude of the procedure, CCRS offers the potential of prolonged survival, or indeed cure, particularly for those diagnosed with PMP. Accumulated 10-year survival rates for 1904 PMP patients after CCRS, in countries including the United Kingdom (UK), indicated survival rates of 74%.

Empirical studies conclude that 'recovery' from the procedure, to preoperative or reference population quality of life scores, across the domains of physical, emotional and psychosocial health, typically occurs 3 - 12 months postoperatively. Notably, however, the dominant paradigm of inquiry adopted in this field is positivist, with survey work accounting for 31/36 of the fully published studies located through a systematic literature search to have examined the impact of CCRS on patients. Such work is limited in its ability to explicate the personal meaning that people may attribute to their lived experience of recovery. Moreover, the remaining five studies have not acquired an understanding of personal meaning over time, across the course of postoperative recovery, in what is likely to be a profound example of postoperative experience with implications beyond those highlighted by positivistic work.

This study aims to fill this gap in the knowledge base by providing a nuanced understanding of the lived experience of recovery over time, from the perspective of patients who have undergone CCRS surgery, with the view to inform future supportive measures for CCRS patients in particular.

There is also a secondary motive for conducting this study.

Recovery is a term used frequently in literature to describe the process that CCRS patients undergo. On occasion, authors insinuate that their study participants (or at least some) experience a complete recovery.

However, the dictionary definition of recovery is 'a return to a normal state of health, mind, or strength', and it is perhaps questionable whether such a definition applies a completely adept description to patients who have experienced CCRS, or indeed any major illness, injury or treatment. Do survivors ever truly recover? Is it not a 'new normal' to some degree? There are increasing reasons to doubt that the definition holds true in such cases, on physical, emotional or psychosocial bases.

For instance, many examples of literature within the field of survivorship following major illness such as cancer, seem to indicate that many survivors continue to experience issues pertaining to their illness, even years after it is diagnosed or treated. Foster et al. (2009) found that 20-30% of survivors, five or more years after their treatment, consistently reported problems associated with cancer and its treatment. Elliott et al. (2011) found in an online survey of 4892 individuals, of whom 780 were cancer survivors, that survivors 'were significantly more likely to report poor[er] health outcomes … than those with no history of cancer or a chronic condition' (p11). These works are quantitative in nature, and it may be that qualitative work, particularly as it increases in number, will highlight further changes that distinguish survivor's lives from their pre-illness lives. Ohlsson-Nevo (2011) for example, lead with the theme that 'life is normal, and yet not' to describe the experiences of colorectal cancer survivors.

Given the potential that many do not experience a recovery in the full sense, Foster and Fenlon (2011) and Horikoshi and Futawatari (2017) speculate that cancer survivor experiences, in particular, are more akin to a process of adaptation such as that necessitated by chronic illness (previously discussed by the 'biographical disruption' work of Bury (1991), Charmaz (1991) Dorsett (1991) and Frank (1997)).

This study provides the opportunity to longitudinally examine patient perceptions of the concept of 'recovery': How do survivors of major illness or treatment define recovery as a term, both as a process and as an outcome? Do such perceptions change over time? Even if they are physically, emotionally or psychosocially 'recovered', do survivors think or live their lives differently as a result of their experiences? In what ways do people not recover? Do they consider themselves as recovered?

In conclusion, this study seeks a longitudinal and detailed understanding of the experience of recovery from CCRS, beyond that currently recognised by empirical work. This will be useful in informing supportive measures for CCRS patients as they 'recover', and furthermore will increase our understanding of recovery as a concept.

The study utilises interpretive phenomenological analysis (IPA) as a methodological framework, which is suitable in meeting such objectives in light of its three core principles. In being phenomenological, this study acknowledges that the study of lived experience is a valid means of understanding the recovery process. It encourages the researcher to suspend their preconceptions as much as possible and to be fully receptive and inquisitive to the experience as it is conveyed. In being hermeneutical, this study acknowledges that researcher-led interpretation is necessary in fully understanding lived experience, particularly in the context of the sensitive timeframe in which the research will be performed, and in bringing to light the temporal changes that may occur as the study progresses. Lastly, in being idiographic, this study recognises that individual lived experiences of recovery following CCRS are likely to be unique and rich, and deserve in-depth consideration. It also acknowledges that literature exists in the field, and that this may be re-evaluated in the light of in-depth findings. An in-depth understanding of the experiences of CCRS patients as they 'recover' from their surgery, and the meanings of 'recovery' to them during this time, should therefore be attained through the use of IPA.

This study will implement a longitudinal interview-based design with sequential data collection points running over an approximate 12-14 month period.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible to be invited to participate in the study if…

1. They are electively booked in…
2. … for Complete Cytoreducive Surgery (CCRS)…
3. … for 'four-quadrant' Pseudomyxoma peritonei (PMP)…
4. … at Basingstoke and North Hampshire Hospital (BNHH).
5. They are 16 years old or over.
6. They live within an approximate 100 mile radius of BNHH.
7. They are able to converse in English, without the assistance of others.
8. They are deemed able to independently make an informed decision whether or not to participate in the study (i.e. the individual must appear able to understand, retain and use or weigh up information as part of decision making processes)

Exclusion Criteria:

1. Potential participants are excluded if they have had a previous diagnosis of cancer.
2. Potential participants are also excluded if they have had, or are due to have, a treatment of systemic chemotherapy.

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Potential participants are likely to be approached at outpatient appointments by clinical nurse specialists.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
To gather an in-depth understanding of the experiences of patients following complete cytoreductive surgery, using interpretative phenomenological analysis | 1 Year
  The primary objective of the study is to elicit an in-depth understanding of the lived experience of 'recovery' in the year following CCRS. Up to ten study participants will be interviewed on up to six occasions, and the data produced will be analysed using interpretative phenomenological analysis.
To gather an in-depth understanding of the meaning of recovery to patients after complete cytoreductive surgery, using interpretative phenomenological analysis | 1 Year
  The secondary objective of the study is to identify the meaning(s) of 'recovery' to study participants over time in the year following CCRS. Up to ten study participants will be interviewed on up to six occasions, and the data produced will be analysed using interpretative phenomenological analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Basingstoke and North Hampshire Hospital, Basingstoke, Hampshire, United Kingdom

REFERENCES:
- [Background] Glehen O, Kwiatkowski F, Sugarbaker PH, Elias D, Levine EA, De Simone M, Barone R, Yonemura Y, Cavaliere F, Quenet F, Gutman M, Tentes AA, Lorimier G, Bernard JL, Bereder JM, Porcheron J, Gomez-Portilla A, Shen P, Deraco M, Rat P. Cytoreductive surgery combined with perioperative intraperitoneal chemotherapy for the management of peritoneal carcinomatosis from colorectal cancer: a multi-institutional study. J Clin Oncol. 2004 Aug 15;22(16):3284-92. doi: 10.1200/JCO.2004.10.012. PMID 15310771
- [Background] Sugarbaker PH. Peritonectomy procedures. Ann Surg. 1995 Jan;221(1):29-42. doi: 10.1097/00000658-199501000-00004. PMID 7826158
- [Background] Chua TC, Yan TD, Saxena A, Morris DL. Should the treatment of peritoneal carcinomatosis by cytoreductive surgery and hyperthermic intraperitoneal chemotherapy still be regarded as a highly morbid procedure?: a systematic review of morbidity and mortality. Ann Surg. 2009 Jun;249(6):900-7. doi: 10.1097/SLA.0b013e3181a45d86. PMID 19474692
- [Background] Dube P, Sideris L, Law C, Mack L, Haase E, Giacomantonio C, Govindarajan A, Krzyzanowska MK, Major P, McConnell Y, Temple W, Younan R, McCart JA. Guidelines on the use of cytoreductive surgery and hyperthermic intraperitoneal chemotherapy in patients with peritoneal surface malignancy arising from colorectal or appendiceal neoplasms. Curr Oncol. 2015 Apr;22(2):e100-12. doi: 10.3747/co.22.2058. PMID 25908915
- [Background] Shan LL, Saxena A, Shan BL, Morris DL. Quality of life after cytoreductive surgery and hyperthermic intra-peritoneal chemotherapy for peritoneal carcinomatosis: A systematic review and meta-analysis. Surg Oncol. 2014 Dec;23(4):199-210. doi: 10.1016/j.suronc.2014.10.002. Epub 2014 Oct 28. PMID 25466850
- [Background] Stearns AT, Malcomson L, Punnett G, Abudeeb H, Aziz O, Selvasekar CR, Fulford PE, Wilson MS, Renehan AG, O'Dwyer ST. Long-term Quality of Life After Cytoreductive Surgery and Heated Intraperitoneal Chemotherapy for Pseudomyxoma Peritonei: A Prospective Longitudinal Study. Ann Surg Oncol. 2018 Apr;25(4):965-973. doi: 10.1245/s10434-017-6326-0. Epub 2018 Jan 8. PMID 29313146
- [Background] Jess P, Iversen LH, Nielsen MB, Hansen F, Laurberg S, Rasmussen PC. Quality of life after cytoreductive surgery plus early intraperitoneal postoperative chemotherapy for pseudomyxoma peritonei: a prospective study. Dis Colon Rectum. 2008 Jun;51(6):868-74. doi: 10.1007/s10350-008-9223-6. Epub 2008 Feb 23. PMID 18297361
- [Background] Seretis C, Youssef H. Quality of life after cytoreductive surgery and intraoperative hyperthermic intraperitoneal chemotherapy for peritoneal surface malignancies: a systematic review. Eur J Surg Oncol. 2014 Dec;40(12):1605-13. doi: 10.1016/j.ejso.2014.08.477. Epub 2014 Sep 6. PMID 25242382
- [Background] Smith JA, Flowers P and Larkin M (2009) IPA Theory, Method and Research. Sage Publications, Great Britain
- [Background] Smith JA (1996) Beyond the divide between cognition and discourse: Using interpretative phenomenological analysis in health psychology. Psychology and health 11(2): 261-71